CLINICAL TRIAL: NCT02777164
Title: Evaluation of a Three Dimensional Functional Metabolic Imaging and Risk Assessment System for Classifying Women at High Risk of Breast Cancer
Brief Title: Evaluation of a 3D Functional Metabolic Imaging and Risk Assessment System for Classifying Women at High Risk of Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision, not safety related
Sponsor: Real Imaging Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 960-CSP-USA_MIRA_USS2
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MIRA device imaging (Experimental): MIRA Device imaging for adjunctive detection of breast cancer
  Interventions: Device: MIRA device imaging

INTERVENTIONS:
Device: MIRA device imaging — MIRA Device imaging for adjunctive detection of breast cancer
  Other Names: Real Imager 8

SUMMARY:
The objective of the study is to estimate the diagnostic accuracy of cancer detection when MIRA technology is combined with mammography, by evaluating the area under the ROC curve (AUC) of mammography vs. mammography plus MIRA. This evaluation will be done in a Reader Study on a subset of women with histology confirmed cancer and healthy women with dense breast.

ELIGIBILITY:
Inclusion Criteria:

A. Subjects who are asymptomatic and scheduled to undergo routine screening mammography

OR

B. Subjects scheduled for image guided needle biopsy as a result of findings obtained during standard of care imaging modalities

AND

C. Subjects has a prior mammogram and have been diagnosed with extremely or heterogeneously dense breast tissue (Density C or D)

Exclusion Criteria:

1. Male by birth.
2. Individual is less than 30 and greater than 70 years old.
3. Contraindication to bilateral mammography or MRI
4. Subjects who are unable to read, understand and execute the informed consent procedure.
5. Subjects who have had mammography ultrasound or MRI examination performed on the day of the study prior to MIRA scan.
6. Subjects who have significant existing breast trauma.
7. Subjects who have undergone lumpectomy/mastectomy.
8. Subjects who have undergone breast reduction or breast augmentation.
9. Subjects who have undergone any other type of breast surgery, excluding surgical biopsy.
10. Subjects who have large breast scar / Breast deformation
11. Subjects who have undergone a breast needle biopsy or a surgical biopsy within the 6 month period prior to their intended enrollment into the study.
12. Subjects who have a temperature > 100° F (37.8C) degrees on the day of the MIRA imaging
13. Subjects who are pregnant or lactating
14. Subjects with known Raynaud's Disease
15. Subjects that are claustrophobic or have physical limitations that do allow them to sit in the system chair for the required imaging session.
16. Subjects with implanted pacemaker/defibrillator, implanted venous access device (portacath) or other implanted devices
17. Subject with kidney failure
18. Subject with known allergy to gadolinium
19. Subject with a history of multiple contrast MRI scans (more than 4 MRI scans over the past two year)
20. Inmates (45 CFR 46.306) or mentally disabled individuals
21. Subjects with a BI-RADS category 6 (e.g. for which mammogram was performed for the purpose of planning cancer therapy)
22. Subjects currently participating in another investigational clinical study
23. Subjects who participated in the Calibration Phase will not be able to participate in the Testing Phase

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 740 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
The difference in the area under the ROC curve (AUC) of mammography plus MIRA compared to mammography alone. | 19 months

CONTACTS AND LOCATIONS:
Overall Officials: David Izhaky, Study Director — Real Imaging Ltd.
Locations (1):
- MemorialCare Breast Center, Saddleback Memorial, Laguna Hills, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's Web site — http://www.realimaging.com/